CLINICAL TRIAL: NCT00218140
Title: Effects of Nicotine Patch in Men and Women
Brief Title: Effectiveness of the Nicotine Patch in Suppressing Nicotine Withdrawal Symptoms in Women Versus Men - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11082-1; R01-11082-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: tobacco
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

INTERVENTIONS:
Drug: nicotine transdermal system

SUMMARY:
Women typically have a more difficult time quitting smoking than men. Little research has been done to understand the differences between men and women that may cause this distinction. This study will assess whether the reduced effectiveness of nicotine replacement therapy in women is caused by gender differences in the withdrawal suppression induced by nicotine replacement therapy.

DETAILED DESCRIPTION:
Smoking can cause a variety of cancers, cardiovascular disorders, and other health problems. Quitting smoking greatly decreases one's risk for these problems. Studies have shown, however, that quitting smoking is more difficult for women than men. Despite that knowledge, little research has been done to try to understand the mechanistic differences between men and women that may cause this distinction. This study will assess whether the reduced effectiveness of nicotine replacement therapy in women is caused by physical and psychological gender differences in the withdrawal suppression induced by nicotine replacement therapy.

Participants in this double-blind study will attend 4 treatment sessions, each approximately 6.5 hours long and each corresponding to one of four transdermal nicotine replacement patch doses (0, 7, 21, or 42 mg). Sessions will be separated by at least 48 hours to avoid carryover effects. Immediately following arrival at each session, participants' expired air carbon monoxide (CO) levels will be measured to verify that the participant has not smoked for at least 8 hours prior to the visit. If the CO level meets the necessary criteria to proceed, a baseline blood sample will be obtained, followed by additional blood samples every 30 minutes. Baseline nicotine withdrawal levels will be assessed using questionnaires. Computerized recordings of physiological responses will also commence and will continue throughout the session. These response measures will include heart rate, percent oxygen saturation, skin temperature, systolic and diastolic blood pressure, and mean arterial pressure. Upon completion of baseline measures, participants will receive a randomly assigned dose of nicotine replacement therapy, in the form of three patches placed on the participants' back. The patches will be removed after 6 hours and the participant will be assessed for any residual effects from the medication.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least 15 cigarettes a day for at least 2 years prior to enrollment
* Has an afternoon carbon monoxide level of at least 15 ppm
* Agree to use an effective form of contraception for the duration of the study

Exclusion Criteria:

* History of chronic health problems
* History of psychiatric conditions
* History of or active cardiovascular disease
* History of or active high or low blood pressure
* History of or active seizure condition
* History of or active peptic ulcers
* History of or active diabetes
* Pregnant
* Score of greater than 17 on the Beck Depression Inventory

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0
Dates: Study Completion 2005-04

PRIMARY OUTCOMES:
Physiological measures
Tobacco withdrawal
Behavioral accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eissenberg, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- University, Richmond, Virginia, United States